CLINICAL TRIAL: NCT07068256
Title: Comparison Between Therapeutic Efficacy of Itraconazole Pulse Therapy and Terbinafine Therapy in Treatment of Tinea Capitis in Pediatric Population.
Brief Title: Efficacy Comparison of Itraconazole Pulse Therapy and Terbinafine Therapy in Treatment of Tinea Capitis in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRSAIMA-JHLAHORE
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Tinea Capitis
MeSH Terms: conditions — Tinea Capitis | interventions — Terbinafine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terbinafine group (Experimental): Patients will be given terbinafine in a dose of 62.5 mg for less than 20 kg body weight, 125 mg from 20 to 40 kg, and 250 mg for more than 40 kg for a period of 4 weeks.
  Interventions: Drug: Terbinafine
- Itraconazole group (Experimental): Patients will receive itraconazole a dose of 5 mg/kg/day for 7 days and then 14 days off. Three such pulses will be given to the patients of this group.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Terbinafine — Terbinafine will be given at a dose of 62.5 mg in patients with a body weight < 20 kg, 125 mg from 20 to 40 kg, and 250 mg in > 40 kg for a period of 4 weeks.
  Arms: Terbinafine group
Drug: Itraconazole — Itraconazole will be given at a dose of 5 mg/kg/day for 7 days and then 14 days off. Three such pulses will be given to the patients.
  Arms: Itraconazole group

SUMMARY:
Several studies globally have assessed the efficacy of terbinafine and itraconazole in the treatment of tinea capitis, but local data in this regard is scarce. Therefore, this study was planned with the aim of assessing the difference between the therapeutic efficacy of itraconazole pulse therapy and terbinafine in children with tinea capitis.

DETAILED DESCRIPTION:
The existing literature carries varying results between the effectiveness of itraconazole pulse therapy and continuous terbinafine therapy in treating tinea capitis, and local data in this regard is also scarce. The findings of this study would not only add to the statistics but would also help clinicians to offer a treatment modality in pediatric tinea capitis, which should have better efficacy, a low incidence of side effects, and better patient compliance.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Aged 1-13 years
* With KOH mount positive before start of treatment
* Duration of disease more than 1 month

Exclusion Criteria:

* KOH mount negative before starting the treatment
* Topical treatment with antifungal agents within past 4 weeks
* Systemic treatment with antifungal agents within past 4 weeks
* Patients with active liver disease
* Patients with elevated liver enzymes

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Fungus eradication | 9 weeks
  Treatment will be labeled efficacious if the patient will be cured clinically as well as mycologically, i.e., samples treated with KOH will show no fungal elements.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Aslam, Principal Investigator — Jinnah Hospital/Allama Iqbal Medical College, Lahore; Fahad Iqbal, FCPS, Study Director — Sir Ganga Ram Hospital Lahore
Locations (1):
- Jinnah Hospital/Allama Iqbal Medical College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request